CLINICAL TRIAL: NCT03747939
Title: A Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Apremilast (CC-10004) in Subjects With Early, Oligoarticular Psoriatic Arthritis Despite Initial Stable Treatment With Either NSAIDS and/or ≤ 1 Conventional Synthetic DMARD
Brief Title: Efficacy, Safety, and Tolerability Study of Apremilast to Treat Early Oligoarticular Psoriatic Arthritis.
Acronym: FOREMOST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSA-013; U1111-1224-0216 (Registry Identifier: WHO); 2018-002735-26 (EudraCT Number)
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Arthritis, Psoriatic
Keywords: Oligoarthritis; PsA; Apremilast; Oral tablet; Background therapy; Standard of care
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apremilast 30 mg twice daily ± NSAIDs, ≤ 1 csDMARD (Experimental): Subjects will take ORAL tables of apremilast for up to 48 weeks (30 mg twice daily). Subjects may also receive stable doses of background therapy (standard or care) with NSAIDs, glucorticosteroids and 1 csDMARD as permitted by protocol. After wk. 24, subjects may change the dose /type of permitted Psoriatic Arthritis medications
  Interventions: Drug: Apremilast (CC-10004)
- Placebo (Placebo Comparator): Subjects will take placebo for up to 24 weeks (twice daily). Subjects may also receive stable doses of background therapy ( standard of care) with NSAIDs, glucocorticosteroids and 1 csDMARD as permitted by protocol. After wk 24, subjects may change the dose /type of permitted PsA medications.
  Interventions: Other: Apremilast (CC-10004) Placebo

INTERVENTIONS:
Drug: Apremilast (CC-10004) — Subjects randomized to apremilast will receive dose-titration for the initial 5 days. Apremilast subjects will receive "dummy" titration at wk. 16 (for early escape subjects) and again at week 24 to maintain the blinding of the original treatment assignments. Investigational product (IP) will be dispensed in blinded dose cards until Week 28. Thereafter, IP will be dispensed in open-label bottles.
  Other Names: Otezla
  Arms: Apremilast 30 mg twice daily ± NSAIDs, ≤ 1 csDMARD
Other: Apremilast (CC-10004) Placebo — Subjects randomized to placebo will receive "dummy" dose-titration for the initial 5 days. Placebo subjects who meet the criteria for early escape at wk. 16 may receive apremilast beginning at wk. 16 and will receive active titration. Remaining placebo subjects will receive active dose titration at week 24. Beginning at wk 24 all subjects will be dispensed active apremilast. Investigational product will be dispensed in blinded dose cards until Week 28. to maintain the blinding of the original treatment assignments. Thereafter, IP will be dispensed in open-label bottles
  Arms: Placebo

SUMMARY:
This clinical study will test the effects of a drug called apremilast in oligoarticular psoriatic arthritis with less than 5 years of disease duration. In previous studies, apremilast has been shown to be safe and efficacious in reducing signs and symptoms of psoriatic arthritis, as well as improving physical function. This study will compare the effects of apremilast to placebo on psoriatic arthritis subjects in which the number of affected joints is limited (greater than 1 but less or equal to 4). About 285 patients worldwide will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 yrs, male or female subject
* Subjects must have signs and symptoms of PsA ≤5 years duration at the time of the Screening Visit
* SJC AND TJC must be >1 and ≤ 4
* For all regions, the local Regulatory Label for treatment with apremilast must be followed.
* Stable doses of protocol-allowed PsA medications
* General good health (except for psoriatic arthritis) as judged by the Investigator, based on medical history, physical examination, and clinical laboratories. (Note: The definition of good health means a subject does not have uncontrolled significant comorbid conditions).
* Comply with protocol-required contraception measures
* Subject meets the Classification Criteria for Psoriatic Arthritis [CASPAR] Criteria for PsA at the Screening visit

Exclusion Criteria:

* Prior use of >2 csDMARD to treat PsA
* Prior exposure to a JAK-inhibitor and/or a biologic DMARD.
* Use of intra-articular (IA) or intra-muscular (IM) glucocorticoid injection within 8 weeks before the Baseline Visit.
* Use of leflunomide within 12 weeks of randomization. Subjects who stopped leflunomide and completed 11 days of treatment with cholestyramine (8 g, 3 x daily) prior to the Baseline Visit may enter the study.
* Prior use of cyclosporine.
* Prior treatment with apremilast, or participation in a clinical study, involving apremilast.
* Use of any investigational drug within 4 weeks of the Baseline Visit, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (114):
- United States (54):
  - Arizona Arthritis and Rheumatology Research, PLLC, Mesa, Arizona
  - Covina Arthritis Clinic, Covina, California
  - Encino Research Center, Encino, California
  - Providence Medical Foundation, Fullerton, California
  - Rheumatology Center of San Diego PC, San Diego, California
  - East Bay Rheumatology Medical, San Leandro, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Robin K Dore MD Inc, Tustin, California
  - Inland Rheumatology Clinical Trials Inc, Upland, California
  - Denver Arthritis Clinic PC, Denver, Colorado
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - Center for Rheumatology, Immunology, and Arthritis, Fort Lauderdale, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Integral Rheumatology and Immunology Specialists, Plantation, Florida
  - Florida Center For Dermatology, Saint Augustine, Florida
  - Clinical Research of West Florida Inc, Tampa, Florida
  - Carol and Frank Morsani Center for Advanced Health Care, Tampa, Florida
  - Baycare Medical Group Inc, Tampa, Florida
  - North Georgia Rheumatology Group PC, Lawrenceville, Georgia
  - RC Rsearch Inc, Hinsdale, Illinois
  - OrthoIllinois, Rockford, Illinois
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Klein and Associates MD, PA - Cumberland, Cumberland, Maryland
  - Klein and Associates MD PA, Hagerstown, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Advanced Rheumatology PC, Lansing, Michigan
  - Arthritis and Rheumatology Center of Michigan, Lansing, Michigan
  - Clinical Research Institute of Michigan, Saint Clair Shores, Michigan
  - Saint Paul Rheumatology PA, Eagan, Minnesota
  - Arthritis, Rheumatic, and Back Disease Associates, Voorhees Township, New Jersey
  - New York University Langone Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Paramount Medical Research and Consulting LLC, Middleburg Heights, Ohio
  - Arthritis and Osteoporosis Center of Southwest Ohio, Middletown, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - West Tennessee Research Institute, llc, Jackson, Tennessee
  - Accurate Clinical Research Incorporated Baytown, Baytown, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Texas Arthritis Center PA, El Paso, Texas
  - West Texas Clinical Research, Lubbock, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - Center for Clinical Studies, Webster, Texas
  - Seattle Rheumatology Associates, Seattle, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
  - West Virginia Research Institute, Morgantown, West Virginia
  - West Virginia Research Institute, South Charleston, West Virginia
- Austria (2):
  - Universitaetsklinikum Allgemeines Krankenhaus Wien Universitaetsklinik fur Innere Medizin I, Vienna
  - Krankenhaus Hietzing, Vienna
- Belgium (4):
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Hopital Erasme, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
  - Ziekenhuis Netwerk Antwerpen Jan Palfijn, Merksem
- Canada (5):
  - Manitoba Clinic, Winnipeg, Manitoba
  - Ottawa Hospital, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Dr Sabeen Anwar Medicine Professional Corporation, Windsor, Ontario
  - Institut de Rhumatologie de Montreal, Montreal, Quebec
- France (4):
  - Centre Hospitalier Regional dOrleans, Orléans
  - Hopital Lariboisiere, Paris
  - Assistance Publique- Hopitaux de Paris AP-HP, Paris
  - CH Toulouse Hopital Pierre-Paul Riquet, Toulouse
- Germany (9):
  - Praxis fur Rheumatologie - Amberg, Amberg
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Service Rheuma Erfurt, Erfurt
  - Klinikum der Johann Wolfgang Goethe-Universitaet Frankfurt/Main, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Rheumazentrum Ruhrgebiet, Herne
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (10):
  - AO Ospedale Policlinico Consorziale Di Bari, Bari
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Universita degli studi Messina, Messina
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Policlinico San Matteo Universita Di Pavia, Pavia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Fondazione Policlinico Tor Vergata, Rome
  - Humanitas Research Hospital Humanitas Mirasole, Rozzano MI
  - Azienda Ospedaliera Universitaria Integrata di Verona Ospedale G B Rossi Borgo Roma, Verona
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - Erasmus Medisch Centrum, Rotterdam
- Russia (10):
  - Kazan State Medical University, Kazan'
  - Kursk Regional Clinical Hospital, Kursk
  - Research Institute of Rheumatology named after V A Nasonova, Moscow
  - Moscow Regional Research Institute n a Vladimirsky, Moscow
  - Research Institute of Clinical and Experimental Lymphology, Novosibirsk
  - Republican Hospital na VA Baranov, Petrozavodsk
  - Municipal Budgetary Healthcare Institution City Emergency Hospital, Rostov-on-Don
  - Mechnikov North-Western State Medical University, Saint Petersburg
  - Medical Center Sanavita, Saint Petersburg
  - Tomsk Regional Clinical Hospital, Tomsk
- Spain (6):
  - Hospital Universitario de Cruces, Barakaldo, Basque Country
  - Hospital Galdakao-Usansolo, Galdakao
  - Hospital Universitario Insular de Gran Canaria, Gran Canaria
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Merida, Mérida
- United Kingdom (8):
  - Royal Berkshire Hospital, Derby
  - Eastbourne District General Hospital, Eastbourne
  - Western General Hospital, Edinburgh Scotland
  - Kings College Hospital, London
  - Luton and Dunstable University Hosptial, Luton
  - Torbay Hospital, Torquay South Devon
  - Royal Cornwall Hospitals Trust, Truro
  - Wolverhampton Road, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Gossec L, Coates LC, Gladman DD, Aelion JA, Vasandani J, Pinter A, Merola JF, Kavanaugh A, Reddy J, Wang R, Brunori M, Klyachkin Y, Deignan C, Mease PJ. Treatment of early oligoarticular psoriatic arthritis with apremilast: primary outcomes at week 16 from the FOREMOST randomised controlled trial. Ann Rheum Dis. 2024 Oct 21;83(11):1480-1488. doi: 10.1136/ard-2024-225833. PMID 39164067
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 80 study centers in Austria, Belgium, Canada, France, Germany, Italy, Spain, the United Kingdom, and the United States from 31 December 2018 to the last participant's last study visit on 05 July 2023.
Pre-assignment Details: Participants with early oligoarticular psoriatic arthritis were randomized in a 2:1 ratio to receive apremilast or placebo. At week 16, participants with no swollen joint count (SJC) improvement could have escaped early to receive apremilast 30 mg BID. At week 24, eligible participants entered the open-label extension phase to receive apremilast 30 mg BID up to week 48. Of the 310 enrolled participants, 2 were enrolled in error and did not receive any dose of investigational product.
Groups:
- Placebo-controlled Phase: Placebo: Participants were randomized to receive placebo twice daily (BID) from day 1. Participants could also have received stable doses of non-steroidal anti-inflammatory drugs (NSAIDs) and 1 conventional synthetic disease-modifying antirheumatic drug (csDMARD).
- Placebo-controlled Phase: Apremilast 30 mg: Participants were randomized to receive apremilast 30 mg BID from day 1. Participants could also have received stable doses of NSAIDs and 1 csDMARD.
- Apremilast-extension Phase: Placebo Then Apremilast 30 mg: Participants were randomized to receive placebo in the placebo-controlled phase, and entered the open-label apremilast-extension phase to receive apremilast 30 mg BID from week 24 to week 48.
- Apremilast-extension Phase: Continued Apremilast 30 mg: Participants were randomized to receive apremilast 30 mg BID in the placebo-controlled phase, and entered the open-label apremilast-extension phase to continue on apremilast 30 mg BID from week 24 to week 48.
Period: Placebo-controlled Phase (Weeks 0 - 24)
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremilast-extension Phase: Placebo Then Apremilast 30 mg | Apremilast-extension Phase: Continued Apremilast 30 mg
Started | 105 | 203 | 0 | 0
Full Analysis Set | 105 | 203 | 0 | 0
Safety Analysis Set (Included participants according to the treatment they actually received.) | 104 | 204 (1 participant randomized to placebo was treated with apremilast.) | 0 | 0
Escaped Early at Week 16 | 24 | 21 | 0 | 0
Completed Week 16 and Continued | 92 | 172 | 0 | 0
Completed (Completed to Week 24 and continued to extension phase) | 87 | 162 | 0 | 0
Not Completed | 18 | 41 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Adverse Event | 8 | 19 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 7 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 7 | 0 | 0
Not completed — Miscellaneous | 0 | 2 | 0 | 0
Period: Apremilast Extension (Weeks 24 - 48)
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremilast-extension Phase: Placebo Then Apremilast 30 mg | Apremilast-extension Phase: Continued Apremilast 30 mg
Started | 0 | 0 | 87 | 162
Received 1 Dose of Investigational Product | 0 | 0 | 86 | 160
Completed | 0 | 0 | 77 | 133
Not Completed | 0 | 0 | 10 | 29
Not completed — Adverse Event | 0 | 0 | 2 | 6
Not completed — Lack of Efficacy | 0 | 0 | 3 | 8
Not completed — Lost to Follow-up | 0 | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 7
Not completed — Other | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Placebo-controlled Phase: Placebo: Participants were randomized to receive placebo BID from day 1. Participants could also have received stable doses of NSAIDs and 1 csDMARD.
- Total: Total of all reporting groups
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Total
Number analyzed (Participants) | 105 | 203 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (13.03) | 51.3 (12.25) | 50.9 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 118 | 169
  Male | 54 | 85 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 1 | 4 | 5
  Black or African American | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 99 | 192 | 291
  Not Collected or Unknown | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 29
  Not Hispanic or Latino | 91 | 185 | 276
  Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Clinical State of Minimal Disease Activity (MDA-Joints) Response at Week 16
Description: MDA is defined as tender joint counts (TJC) ≤ 1 and SJC ≤ 1 plus 3 of the following 5 criteria:
  1. psoriasis body surface area (BSA) ≤ 3%
  2. patient's pain visual analogue scale (VAS) on a 100 mm scale ≤ 15; where 0 indicates 'no pain' and 100 indicates 'pain as severe as can be imagined'
  3. patient's global assessment of disease activity on a 100 mm scale ≤ 20, where 0 represents the lowest level of disease activity and 100 represents the highest.
  4. physical function assessed by Health Assessment Questionnaire Disability Index (HAQ-DI) ≤ 0.5; where 0 represents normal or no difficulty and 3 represents an inability to perform
  5. enthesitis count ≤ 1 based on the Leeds Enthesitis Index; where 0 means nontender and 6 indicates 6 tender tendon insertions.
Time Frame: Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
percentage of participants | 16.0 | 33.9
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Adjusted difference in proportions is the weighted average of the treatment differences across strata formed by two stratification factors, prior/concomitant use of csDMARD and baseline glucocorticosteroid use per Interactive Web Response System (IWRS) data, using Cochran-Mantel-Haenszel (CMH) weights. Two-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel; Two-sided p-value adjusted for prior/concomitant use of csDMARD and baseline glucocorticosteroid use, normalized via Wilson-Hilferty transformation; Adjusted difference in proportions = 18.5, 95% CI 2-sided [8.9 to 28.1] — Apremilast - Placebo

2. Secondary Outcome: Percentage of Participants Who Achieved Remission or Low Disease Activity at Week 16 Based on Clinical Activity in Psoriatic Arthritis (cDAPSA)
Description: The cDAPSA score is based on the numerical summation of 4 disease activity variables: tender and swollen joints, patient's global assessments of disease activity and assessment of pain (VAS). The cDAPSA score ranges from 0 to 154, with a higher score indicating more disease activity.
  cDAPSA remission is defined as a DAPSA score ≤ 4 and low disease activity is defined as a cDAPSA score > 4 but ≤ 13).
Time Frame: Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
percentage of participants | 51.8 | 70.2
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Adjusted difference in proportions is the weighted average of the treatment differences across strata formed by two stratification factors, prior/concomitant use of csDMARD and baseline glucocorticosteroid use per IWRS data, using CMH weights. Two-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted difference in proportions = 18.6, 95% CI 2-sided [7.0 to 30.2] — Apremilast - Placebo

3. Secondary Outcome: Percentage of Participants With SJC ≤ 1 at Week 16
Description: The SJC was based on 66 joints and at week 16 is based on the sentinel joints (i.e., the joints that were affected at baseline). A SJC response is defined as a count ≤ 1.
Time Frame: Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
percentage of participants | 69.0 | 74.0
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3539, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted difference in proportions = 5.1, 95% CI 2-sided [-5.8 to 16.0] — Apremilast - Placebo

4. Secondary Outcome: Percentage of Participants With TJC ≤ 1 at Week 16
Description: The TJC was based on 68 joints and at week 16 was based on the sentinel joints (i.e., the joints that were affected at baseline). A TJC response is defined as a count ≤ 1.
Time Frame: Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
percentage of participants | 44.4 | 66.2
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted difference in proportions = 22.1, 95% CI 2-sided [10.4 to 33.7] — Apremilast - Placebo

5. Secondary Outcome: Percentage of Participants With Patient's Global Assessments of Disease Activity Score of ≤ 20 mm in the VAS at Week 16
Description: The Patient's Global Assessments of Disease Activity is an assessment of how active a participant's psoriatic arthritis was on average during the last week. It was assessed on a VAS ranging from 0 to 100 mm, with a higher score indicating more disease activity. A response is defined as a score ≤ 20 mm.
Time Frame: Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
percentage of participants | 19.1 | 30.4
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0286, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted difference in proportions = 11.8, 95% CI 2-sided [1.7 to 22.0] — Apremilast - Placebo

6. Secondary Outcome: Percentage of Participants With an Assessment of Pain Score ≤ 15 mm in VAS at Week 16
Description: The Patients Pain VAS is the participant's assessment of how much pain they had, on average, during the last week in their joints due to psoriatic arthritis. The VAS score ranges from 0 to 100 mm, with a higher score indicating more pain.
Time Frame: Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
percentage of participants | 13.1 | 29.4
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted difference in proportions = 16.3, 95% CI 2-sided [6.9 to 25.8] — Apremilast - Placebo

7. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Impact of Disease 12-item for Clinical Trials (PsAID-12) Questionnaire Score at Week 16
Description: The PsAID-12 Questionnaire is a 12-item, self-administered questionnaire that reflects the impact of psoriatic arthritis from the perspective of the participant. The overall score ranges from 0 (best status) to 10 (worst status), with a cut-off ≤ 4 representing patient-acceptable symptom state. Analysis was based on a mixed-effects model for repeated measures (MMRM), which included treatment group, time, treatment group by time interaction, prior/concomitant use of csDMARD (naive, prior use only, both prior and concomitant use) and baseline glucocorticosteroid use (yes/no) per IWRS data as factors, and baseline value as a covariate.
Time Frame: Baseline and Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
score on a scale | -0.42 (0.216) | -1.45 (0.178)
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Difference in LS means is based MMRM of the change from baseline; Test type: Superiority; p < 0.0001, MMRM; Difference in LS means = -1.03, 95% CI 2-sided [-1.48 to -0.59] — Apremilast - Placebo

8. Secondary Outcome: Percentage of Participants With a Good or Moderate Psoriatic Arthritis Disease Activity (PASDAS) Score at Week 16
Description: The PASDAS is a weighted index comprising assessments of joints, function, acute-phase response, quality of life, and patient and physician VAS. The score range of the PASDAS is 0 - 10, with worse disease activity represented by higher scores. A good response is defined as a PASDAS score of ≤ 3.2 with improvement from baseline ≥ 1.6 points. A moderate response is defined as a PASDAS score > 3.2 with improvement from baseline ≥ 1.6 points; or PASDAS score < 5.4 with improvement from baseline ≥ 0.8 but < 1.6 points.
Time Frame: Baseline and Week 16
Population: The full analysis set included all participants who were randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 105 | 203
percentage of participants | 42.7 | 59.9
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0043, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted difference in proportions = 17.7, 95% CI 2-sided [5.7 to 29.7] — Apremilast - Placebo

ADVERSE EVENTS:
Time Frame: Week 0 up to week 48 (end of extension phase), and a 4-week observational follow-up (up to 52 weeks).
Description: The safety analysis set included all participants who received at least 1 dose of study medication. For the placebo-controlled phase, participants were included in the treatment group for the treatment they actually received.
Groups:
- Apremilast-exposure: Apremilast 30 mg During Placebo-controlled and Extension Phases: All participants who received apremilast 30 mg BID during the study, including: participants who were randomized to placebo during the placebo-controlled phase, and received apremilast 30 mg during the extension phase; and all participants who received apremilast 30 mg BID during the placebo-controlled phase.
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremilast-exposure: Apremilast 30 mg During Placebo-controlled and Extension Phases
All-Cause Mortality (participants affected / at risk) | 0/104 | 2/204 | 2/291
Serious Adverse Events (participants affected / at risk) | 6/104 | 9/204 | 15/291
Other Adverse Events (participants affected / at risk) | 18/104 | 72/204 | 103/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=104) | Placebo-controlled Phase: Apremilast 30 mg (N=204) | Apremilast-exposure: Apremilast 30 mg During Placebo-controlled and Extension Phases (N=291)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Troponin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=104) | Placebo-controlled Phase: Apremilast 30 mg (N=204) | Apremilast-exposure: Apremilast 30 mg During Placebo-controlled and Extension Phases (N=291)
Diarrhoea (Gastrointestinal disorders) | 11 | 47 | 69
Nausea (Gastrointestinal disorders) | 4 | 22 | 28
COVID-19 (Infections and infestations) | 3 | 7 | 19
Headache (Nervous system disorders) | 3 | 16 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03747939/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03747939/SAP_001.pdf